CLINICAL TRIAL: NCT05550688
Title: The Effect of Weight Gain After Smoking Cessation Increased the Risk of Type 2 Diabetes in Individuals With Nonalcoholic Fatty Liver Disease
Brief Title: Weight Gain After Smoking Cessation and NAFLD
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NAFLD_quitsmoking
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Nonalcoholic Fatty Liver Disease; Type 2 Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NAFLD and NAFLD-free cohort: The investigators diagnosed nonalcoholic fatty liver based on abdominal ultrasonography and ruled out excessive alcohol consumption and other etiologies of liver disease according to the Chinese Liver Disease Association.

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is rapidly becoming the most common chronic liver disease. Considering that there are no approved pharmacological treatments, lifestyle modification is necessary and challenging to reduce the risk of type 2 diabetes mellitus (T2DM) in patients with NAFLD.

Cigarette smoking has a significant negative impact on public health, causing more than 480,000 deaths each year. Smoking has been reported as a risk factor for NAFLD and might accelerate liver disease progression. Therefore, it is recommended that patients with NAFLD quit smoking. However, smoking cessation could be complicated by weight gain. Thus, it is important to assess the impact of weight change after smoking cessation on patients with NAFLD. Proper management of post-cessation weight could maximize its health benefits.

In this large-scale cohort study, the investigators aimed to assess the effects of smoking cessation and subsequent weight change on risks of incident T2DM in individuals with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

(i) age>=18 years.

Exclusion Criteria:

(i) with missing information on ultrasound, smoking status, and weight; (ii) with excess alcohol intake or history of chronic liver disease at baseline; (iii) female subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators enrolled participants who took annual health examinations at Zhenhai Lianhua Hospital in 2007.
Sampling Method: Non-Probability Sample
Enrollment: 12941 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Weight Change after smoking cessation on incident T2DM in NAFLD individuals | a 7-year cohort study
  The investigators used Cox proportional hazard models to estimate hazard ratios (HRs) and 95% CIs for the associations of weight change during smoking cessation with the incidence of T2DM. The investigators did not find any evidence of violation of the proportional hazard assumption. In multivariable models, the investigators constructed three nested models for analysis: (i) model 1 adjusted for age, and body mass index; (ii) model 2, model 1 plus drinking status; (iii) model 3, model 2 plus aspartate aminotransferase, total cholesterol, triacylglycerol, creatinine, albumin, and systolic blood pressure.
Weight Change after smoking cessation on incident T2DM in NAFLD-free individuals | a 7-year cohort study
  The investigators used Cox proportional hazard models to estimate hazard ratios (HRs) and 95% CIs for the associations of weight change during smoking cessation with the incidence of T2DM. The investigators did not find any evidence of violation of the proportional hazard assumption. In multivariable models, the investigators constructed three nested models for analysis: (i) model 1 adjusted for age, and body mass index; (ii) model 2, model 1 plus drinking status; (iii) model 3, model 2 plus aspartate aminotransferase, total cholesterol, triacylglycerol, creatinine, albumin, and systolic blood pressure.

SECONDARY OUTCOMES:
Mediation analysis of smoking relapse on incident T2DM | a 7-year cohort study
  The investigators conducted a mediation analysis to assess whether the association between smoking status and NAFLD was mediated by smoking relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China